CLINICAL TRIAL: NCT01733797
Title: Randomised Pilot Study of Therabite® Versus Wooden Spatula in the Amelioration of Trismus in Head and Neck Cancer Patients. (Trismus Trial)
Brief Title: Trismus Trial of Therabite vs Wooden Spatula in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brynn Chappell (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Brynn Chappell, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09DOG0843; ISRCTN79084153 (Registry Identifier: ISRCTN); PB-PG-0610-22317 (Other Grant/Funding Number: NIHR Research for Patient Benefit)
Record Dates: First submitted 2012-11-19; First posted 2012-11-27 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Oropharyngeal Cancer; Oral Cancer
Keywords: Trismus; Therabite; Wooden spatula; Head and Neck cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Mouth Neoplasms; Trismus; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wooden spatula (Experimental)
  Interventions: Device: Wooden spatula
- Therabite (Experimental)
  Interventions: Device: Therabite

INTERVENTIONS:
Device: Wooden spatula — Lollipop sticks placed between incisors
  Arms: Wooden spatula
Device: Therabite — Hand held device placed in mouth that exercises the jaw
  Arms: Therabite

SUMMARY:
The trial will compare exercises using Therabite® versus wooden spatulas to prevent or relieve trismus in patients with stage 3 and 4 oral/oropharyngeal cancer.

DETAILED DESCRIPTION:
Trismus is defined as a tightening of jaw opening. The negative impact of Trismus on the quality of life of head and neck cancer patients is well established. It affects eating, drinking, speaking and social function and is often as debilitating as any disfigurement resulting from treatment.

The use of jaw exercises using a Therabite appliance following treatment has been shown to reduce the level of Trismus in small studies. Many UK centres, however, use stacked wooden spatulas inserted between the incisors as a means of passive exercise. There is anecdotal evidence that suggests the use of exercises prior to treatment may help reduce the severity of the Trismus experienced by the patient.

This study will enrol 112 head and neck cancer patients allocated by chance to use either the Therabite or wooden spatula and patients will be asked to perform mouth exercises on a daily basis for 6 months.

There is a need to evaluate both the clinical effectiveness and cost-effectiveness of Therabite as opposed to wooden spatulas to determine whether they should be adopted as standard care in head and neck cancer patients.

In this pilot trial, the investigators will measure benefits of Therabite to patients, as compared to usual care with wooden spatulas. Mouth opening will be the key outcome for the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written informed consent
* Aged 18 years and older
* Able to read and write English sufficiently to be able to complete questionnaires
* Stage 3/4 oral and oropharyngeal cancer patients undergoing:

Primary chemoradiotherapy or Surgical free flap plus post operative radiotherapy or post operative chemoradiotherapy

* All patients will receive 60-70 Gy in 30-35 fractions over 6 to 7 weeks to the region of the pterygoid muscles.
* All patients will have at least some trismus as indicated by subjective tightening in the jaw.

Exclusion Criteria:

* <12mm mouth opening (cannot use Therabite)
* Anatomically unable to use Therabite for example patients who may only be partially dentate and to use the Therabite would place extreme stress on the existing teeth
* Cognitive impairment as judged by the clinicians
* International patients treated who will not have routine UK follow up.
* Previous surgery or RT to the head and neck prior to this diagnosis
* Any patient who has no subjective tightening of the jaw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Jaw measurement | Baseline, 3 months and 6 months at hopsital
  Willis bite calliper will be used to measure the jaw opening at baseline, 3 and 6 months

SECONDARY OUTCOMES:
Adherence to intervention | up to 6 months
  Adherence to device use will be captured by the patient on a progress log
Quality of Life | Baseline, 3 and 6 months
Health economic analysis | Baseline, 3 and 6 months
  Patients hospital and service use will be captured at Baseline, 3 and 6 months during interviews with the patient.
  Units used will be days in hospital or number of appointments

CONTACTS AND LOCATIONS:
Overall Officials: Prof Slevin, Study Chair — The Christie NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Queen Victoria Hospital, East Grinstead
  - Aintree University Hospitals NHS Foundation Trust, Liverpool
  - The Christie NHS Foundation Trust, Manchester
  - York Hospital, York

REFERENCES:
- [Derived] Lee R, Molassiotis A, Rogers SN, Edwards RT, Ryder D, Slevin N. Protocol for the trismus trial-therabite versus wooden spatula in the amelioration of trismus in patients with head and neck cancer: randomised pilot study. BMJ Open. 2018 Mar 30;8(3):e021938. doi: 10.1136/bmjopen-2018-021938. PMID 29602860
- [Derived] Lee R, Yeo ST, Rogers SN, Caress AL, Molassiotis A, Ryder D, Sanghera P, Lunt C, Scott B, Keeley P, Edwards RT, Slevin N. Randomised feasibility study to compare the use of Therabite(R) with wooden spatulas to relieve and prevent trismus in patients with cancer of the head and neck. Br J Oral Maxillofac Surg. 2018 May;56(4):283-291. doi: 10.1016/j.bjoms.2018.02.012. Epub 2018 Mar 9. PMID 29526341
- See also: Christie NHS website — http://www.christie.nhs.uk/